CLINICAL TRIAL: NCT02164539
Title: 200699: A Clinical Study to Evaluate Four Doses of Umeclidinium Bromide in Combination With Fluticasone Furoate in COPD Subjects With an Asthmatic Component
Brief Title: Evaluation of Umeclidinium Bromide in Combination With Fluticasone Furoate in COPD Subjects With an Asthmatic Component
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 200699
Record Dates: First submitted 2014-06-12; First posted 2014-06-16 (Estimated); Results first posted 2016-06-28 (Estimated); Last update posted 2017-10-11 (Actual); Status verified 2017-10

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: GSK573719; asthma; UMEC; FF; GSK2829332; persistent obstruction; GW685698; Fluticasone Furoate; COPD; umeclidinium bromide
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment Phase A (Experimental): Eligible subjects will enter a 4-week run-in period and will receive fluticasone propionate/salmeterol. Subjects will then be randomized to receive fluticasone furoate 100 mcg, fluticasone furoate/umeclidinium bromide 100/15.6 mcg, fluticasone furoate/umeclidinium bromide 100/62.5 mcg, fluticasone furoate/umeclidinium bromide 100/125 mcg, fluticasone furoate/umeclidinium bromide 100/250 mcg, or fluticasone furoate/vilanterol 100/25 mcg, respectively for 4 weeks
  Interventions: Drug: FF; Drug: UMEC; Drug: VI
- Treatment Phase B (Experimental): Subjects completing Treatment Phase A will be randomized to receive either fluticasone furoate/umeclidinium bromide100/250 mcg or fluticasone furoate/umeclidinium bromide/vilanterol 100/250/25 mcg for 1 week.
  Interventions: Drug: FF; Drug: UMEC; Drug: VI
- Treatment Phase C (Experimental): Subjects completing Treatment Phase B will be randomized to receive either the same treatment as in Treatment Phase B, or the same treatment minus the umeclidinium bromide component, for 1 week.
  Interventions: Drug: FF; Drug: UMEC; Drug: VI

INTERVENTIONS:
Drug: FF — Fluticasone furoate is available as fluticasone furoate inhalation powder (100 mcg per blister), combination of fluticasone furoate/umeclidinium bromide inhalation powder (fluticasone furoate: 100 mcg per blister, umeclidinium bromide: 15.6, 62.5, 125, or 250 mcg per blister) and combination of fluticasone furoate/vilanterol inhalation powder (fluticasone furoate: 100 mcg per blister, vilanterol: 25 mcg per blister)
Drug: UMEC — Umeclidinium bromide is available as combination of fluticasone furoate/umeclidinium bromide inhalation powder (fluticasone furoate: 100 mcg per blister, umeclidinium bromide: 15.6, 62.5, 125, or 250 mcg per blister)
Drug: VI — Vilanterol is available as vilanterol inhalation powder (25 mcg per blister) and combination of fluticasone furoate/vilanterol inhalation powder (fluticasone furoate: 100 mcg per blister, vilanterol: 25 mcg per blister)

SUMMARY:
The purpose of this study is to evaluate the dose-response of 4 doses of umeclidinium bromide in combination with fluticasone furoate compared with fluticasone furoate monotherapy in chronic obstructive pulmonary disease participants with an asthmatic component. The fluticasone furoate/umeclidinium bromide treatments will also be compared to the once-daily inhaled corticosteroid/long-acting beta agonist combination fluticasone furoate/vilanterol.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* COPD with evidence of an asthmatic component as demonstrated by spirometry, reversibility and current therapy at screening as follows:

  * Post-bronchodilator morning (AM) FEV1 >=50% and <=80% of the predicted normal value at Visit 1
  * Pre- and post-bronchodilator FEV1/FVC ratio <0.7.
  * Demonstrated reversibility by >=12% and >=200 mL increase in FEV1 following albuterol at Visit 1.
  * A need for regular controller therapy (i.e., inhaled corticosteroids alone or in combination with a long-acting beta-agonist or leukotriene modifier, etc.) for a minimum of 12 weeks prior to Visit 1.
* Outpatient subjects who are smokers or non-smokers.

Exclusion Criteria:

* History of life-threatening respiratory event within the last 5 years.
* Unresolved respiratory infection
* Recent Severe COPD or Asthma Exacerbation
* Risk factors for pneumonia
* Hospitalization for pneumonia within 3 months
* Concurrent respiratory disease other than chronic obstructive pulmonary disease or asthma.
* Other uncontrolled condition or disease state that, in the opinion of the investigator, would put the safety of the subject at risk through study participation or would confound the interpretation of the efficacy results if the condition/disease exacerbated during the study.
* Viral hepatitis or HIV
* Current or chronic history of liver disease, known hepatic or biliary abnormalities
* Drug or milk protein allergy
* Administration of prescription or over-the-counter medication that would significantly affect the course of COPD or asthma, or interact with study drug
* Subjects with lung volume reduction surgery within 12 months prior to screening.
* Use of long-term oxygen therapy (LTOT)
* Requirement for nebulized therapy
* Participation in the acute phase of a pulmonary rehabilitation program within 4 weeks
* Unstable or life-threatening cardiac disease
* Abnormal and clinically significant 12-Lead Electrocardiogram (ECG) finding
* Diseases preventing the use of anticholinergics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 338 (Actual)
Dates: Start 2014-07-01; Primary Completion 2015-07-01 (Actual); Study Completion 2015-07-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (54):
- United States (14):
  - GSK Investigational Site, Newport Beach, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Upland, California
  - GSK Investigational Site, Sunset, Louisiana
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Medford, Oregon
  - GSK Investigational Site, Gaffney, South Carolina
  - GSK Investigational Site, Greenville, South Carolina
  - GSK Investigational Site, Rock Hill, South Carolina
  - GSK Investigational Site, Spartanburg, South Carolina
  - GSK Investigational Site, Union, South Carolina
  - GSK Investigational Site, Morgantown, West Virginia
- Argentina (7):
  - GSK Investigational Site, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - GSK Investigational Site, San Rafael, Mendoza Province
  - GSK Investigational Site, Rosario, Santa Fe Province
  - GSK Investigational Site, San Miguel de Tucumán, Tucumán Province
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Mendoza
  - GSK Investigational Site, San Miguel de Tucumán
- Germany (7):
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Neu-Isenburg, Hesse
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Leipzg, Saxony
  - GSK Investigational Site, Teuchern, Saxony-Anhalt
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg
- Poland (8):
  - GSK Investigational Site, Bialystok
  - GSK Investigational Site, Katowice
  - GSK Investigational Site, Kielce
  - GSK Investigational Site, Lodz
  - GSK Investigational Site, Poznan
  - GSK Investigational Site, Sopot
  - GSK Investigational Site, Zgierz
  - GSK Investigational Site, Żnin
- Romania (8):
  - GSK Investigational Site, Bacau
  - GSK Investigational Site, Bucharest
  - GSK Investigational Site, Cluj-Napoca
  - GSK Investigational Site, Comuna Alexandru Cel Bun
  - GSK Investigational Site, Craiova
  - GSK Investigational Site, Piteşti
  - GSK Investigational Site, Ploieşti
  - GSK Investigational Site, Timișoara
- Russia (6):
  - GSK Investigational Site, Blagoveshchensk
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Nizhny Novgorod
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Saratov
  - GSK Investigational Site, Sestroretsk
- Ukraine (4):
  - GSK Investigational Site, Dnipropetrovsk
  - GSK Investigational Site, Kharkiv
  - GSK Investigational Site, Kiev
  - GSK Investigational Site, Kyiv

REFERENCES:
- [Derived] Lee L, Kerwin E, Collison K, Nelsen L, Wu W, Yang S, Pascoe S. The effect of umeclidinium on lung function and symptoms in patients with fixed airflow obstruction and reversibility to salbutamol: A randomised, 3-phase study. Respir Med. 2017 Oct;131:148-157. doi: 10.1016/j.rmed.2017.08.013. Epub 2017 Aug 14. PMID 28947022

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants (par.) with sufficient signs and symptoms to diagnose as having chronic obstructive pulmonary disease (COPD) and evidence of an asthmatic component as demonstrated by spirometry, reversibility and current therapy at the point of screening were eligible for participation in the study.
Pre-assignment Details: Participants on inhaled corticosteroid therapy over the previous 12 weeks, including a stable dose during the 4 weeks prior to Visit 0, entered the 4-week run-in period on open-label fluticasone propionate 250 microgram (µg) and salmeterol 50 µg combination. Eligible par. were stratified by smoking status, age and randomized to Treatment Phase A.
Groups:
- FF 100 µg: Participants received fluticasone furoate (FF) 100 µg once daily in the morning by inhalation using a dry powder inhaler (DPI) for 4 weeks during Treatment Phase A and 1 week during Treatment Phase C. In addition, all participants received supplemental albuterol/salbutamol via metered-dose inhaler (MDI) to be used on an as-needed basis (rescue medication) throughout the study.
- FF/UMEC 100/15.6 µg: Participants received FF 100 µg in combination with umeclidinium bromide (UMEC) 15.6 µg once daily in the morning by inhalation using a DPI for 4 weeks during Treatment Phase A. In addition, all participants received supplemental albuterol/salbutamol via MDI to be used on an as-needed basis (rescue medication) throughout the study.
- FF/UMEC 100/62.5 µg: Participants received FF 100 µg in combination with UMEC 62.5 µg once daily in the morning by inhalation using a DPI for 4 weeks during Treatment Phase A. In addition, all participants received supplemental albuterol/salbutamol via MDI to be used on an as-needed basis (rescue medication) throughout the study.
- FF/UMEC 100/125 µg: Participants received FF 100 µg in combination with UMEC 125 µg once daily in the morning by inhalation using a DPI for 4 weeks during Treatment Phase A. In addition, all participants received supplemental albuterol/salbutamol via MDI to be used on an as-needed basis (rescue medication) throughout the study.
- FF/UMEC 100/250 µg: Participants received FF 100 µg in combination with UMEC 250 µg once daily in the morning by inhalation using a DPI for 4 weeks during Treatment Phase A and 1 week during Treatment Phase B and C. In addition, all participants received supplemental albuterol/salbutamol via MDI to be used on an as-needed basis (rescue medication) throughout the study.
- FF/VI 100/25 µg: Participants received FF 100 µg in combination with vilanterol trifenatate (VI) 25 µg once daily in the morning by inhalation using a DPI for 4 weeks during Treatment Phase A and 1 week during Treatment Phase C. In addition, all participants received supplemental albuterol/salbutamol via MDI to be used on an as-needed basis (rescue medication) throughout the study.
- FF/UMEC/VI 100/250/25 µg: Participants received FF 100 µg in combination with umeclidinium bromide (UMEC) 250 µg and VI 25 µg once daily in the morning by inhalation using two separate DPIs (FF/UMEC 100/250 & VI 25) for 1 week during Treatment Phase B and C. In addition, all participants received supplemental albuterol/salbutamol via MDI to be used on an as-needed basis (rescue medication) throughout the study.
Period: Treatment Phase A (4 Weeks)
Arm/Group | FF 100 µg | FF/UMEC 100/15.6 µg | FF/UMEC 100/62.5 µg | FF/UMEC 100/125 µg | FF/UMEC 100/250 µg | FF/VI 100/25 µg | FF/UMEC/VI 100/250/25 µg
Started | 41 | 42 | 40 | 46 | 85 | 84 | 0
Completed | 39 | 42 | 39 | 44 | 82 | 83 | 0
Not Completed | 2 | 0 | 1 | 2 | 3 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 1 | 2 | 3 | 1 | 0
Period: Treatment Phase B (1 Week)
Arm/Group | FF 100 µg | FF/UMEC 100/15.6 µg | FF/UMEC 100/62.5 µg | FF/UMEC 100/125 µg | FF/UMEC 100/250 µg | FF/VI 100/25 µg | FF/UMEC/VI 100/250/25 µg
Started | 0 | 0 | 0 | 0 | 166 | 0 | 163
Completed | 0 | 0 | 0 | 0 | 163 | 0 | 162
Not Completed | 0 | 0 | 0 | 0 | 3 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 2 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1 | 0 | 1
Period: Treatment Phase C (1 Week)
Arm/Group | FF 100 µg | FF/UMEC 100/15.6 µg | FF/UMEC 100/62.5 µg | FF/UMEC 100/125 µg | FF/UMEC 100/250 µg | FF/VI 100/25 µg | FF/UMEC/VI 100/250/25 µg
Started | 79 | 0 | 0 | 0 | 84 | 82 | 80
Completed | 78 | 0 | 0 | 0 | 84 | 82 | 78
Not Completed | 1 | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- FF 100 µg: Participants received FF 100 µg once daily in the morning by inhalation using a DPI for 4 weeks in Treatment Phase A. In addition, all participants received supplemental albuterol/salbutamol via MDI to be used on an as-needed basis (rescue medication) throughout the study.
- FF/UMEC 100/15.6 µg: Participants received FF 100 µg in combination with UMEC 15.6 µg once daily in the morning by inhalation using a DPI for 4 weeks in Treatment Phase A. In addition, all participants received supplemental albuterol/salbutamol via MDI to be used on an as-needed basis (rescue medication) throughout the study.
- FF/UMEC 100/62.5 µg: Participants received FF 100 µg in combination with UMEC 62.5 µg once daily in the morning by inhalation using a DPI for 4 weeks in Treatment Phase A. In addition, all participants received supplemental albuterol/salbutamol via MDI to be used on an as-needed basis (rescue medication) throughout the study.
- FF/UMEC 100/125 µg: Participants received FF 100 µg in combination with UMEC 125 µg once daily in the morning by inhalation using a DPI for 4 weeks in Treatment Phase A. In addition, all participants received supplemental albuterol/salbutamol via MDI to be used on an as-needed basis (rescue medication) throughout the study.
- FF/UMEC 100/250 µg: Participants received FF 100 µg in combination with UMEC 250 µg once daily in the morning by inhalation using a DPI for 4 weeks in Treatment Phase A. In addition, all participants received supplemental albuterol/salbutamol via MDI to be used on an as-needed basis (rescue medication) throughout the study.
- FF/VI 100/25 µg: Participants received FF 100 µg in combination with VI 25 µg once daily in the morning by inhalation using a DPI for 4 weeks in Treatment Phase A. In addition, all participants received supplemental albuterol/salbutamol via MDI to be used on an as-needed basis (rescue medication) throughout the study.
- Total: Total of all reporting groups
Arm/Group | FF 100 µg | FF/UMEC 100/15.6 µg | FF/UMEC 100/62.5 µg | FF/UMEC 100/125 µg | FF/UMEC 100/250 µg | FF/VI 100/25 µg | Total
Number analyzed (Participants) | 41 | 42 | 40 | 46 | 85 | 84 | 338
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.4 (8.59) | 55.5 (11.33) | 56.7 (10.14) | 58.2 (10.47) | 57.8 (11.03) | 57.6 (10.95) | 57.5 (10.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 23 | 19 | 18 | 38 | 41 | 160
  Male | 20 | 19 | 21 | 28 | 47 | 43 | 178
Race/Ethnicity, Customized [Number; unit: Participants]
  African American/African Heritage | 1 | 0 | 1 | 1 | 3 | 1 | 7
  White- Arabic/ North African Heritage | 0 | 0 | 0 | 1 | 0 | 0 | 1
  White- White/Caucasian/European Heritage | 40 | 42 | 39 | 44 | 81 | 83 | 329
  Mixed Race | 0 | 0 | 0 | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Clinic Trough Forced Expiratory Volume in One Second (FEV1) at the End of Treatment Phase A (Visit 6/Day 29)
Description: FEV1 is defined as forced expiratory volume in one second and measured in the morning at Visits 1 through 8 between 6:00 and 11:00 electronically by spirometry. Change from Baseline in trough FEV1 is defined as the difference in the value obtained at Visit 6 (24 hours post-dose on Visit 5) and the last acceptable/borderline acceptable value obtained prior to randomization (from Visit 2 pre-bronchodilator or Visit 3 pre-dose). Trough FEV1 is defined as the acceptable/borderline acceptable FEV1 value obtained at Visit 6, approximately 24 hours after morning dosing on Visit 5. ITT population is comprised of all participants randomized to treatment who received at least one dose of randomized study medication in the treatment period. All comparisons for statistical purposes are with the FF 100 µg arm.
Time Frame: Baseline and Day 29
Population: ITT Population. Only those participants available at the specified time point were analyzed.
Measure: Mean (Standard Deviation); unit: Liters
Groups:
- FF 100 µg: Participants received fluticasone furoate (FF) 100 µg once daily in the morning by inhalation using a dry powder inhaler (DPI) for 4 weeks. In addition, all participants received supplemental albuterol/salbutamol via metered-dose inhaler (MDI) to be used on an as-needed basis (rescue medication) throughout the study.
- FF/UMEC 100/15.6 µg: Participants received FF 100 µg in combination with umeclidinium bromide (UMEC) 15.6 µg once daily in the morning by inhalation using a DPI for 4 weeks. In addition, all participants received supplemental albuterol/salbutamol via MDI to be used on an as-needed basis (rescue medication) throughout the study.
- FF/UMEC 100/62.5 µg: Participants received FF 100 µg in combination with UMEC 62.5 µg once daily in the morning by inhalation using a DPI for 4 weeks. In addition, all participants received supplemental albuterol/salbutamol via MDI to be used on an as-needed basis (rescue medication) throughout the study.
- FF/UMEC 100/125 µg: Participants received FF 100 µg in combination with UMEC 125 µg once daily in the morning by inhalation using a DPI for 4 weeks. In addition, all participants received supplemental albuterol/salbutamol via MDI to be used on an as-needed basis (rescue medication) throughout the study.
- FF/UMEC 100/250 µg: Participants received FF 100 µg in combination with UMEC 250 µg once daily in the morning by inhalation using a DPI for 4 weeks. In addition, all participants received supplemental albuterol/salbutamol via MDI to be used on an as-needed basis (rescue medication) throughout the study.
- FF/VI 100/25 µg: Participants received FF 100 µg in combination with vilanterol trifenatate (VI) 25 µg once daily in the morning by inhalation using a DPI for 4 weeks. In addition, all participants received supplemental albuterol/salbutamol via MDI to be used on an as-needed basis (rescue medication) throughout the study.
Arm/Group | FF 100 µg | FF/UMEC 100/15.6 µg | FF/UMEC 100/62.5 µg | FF/UMEC 100/125 µg | FF/UMEC 100/250 µg | FF/VI 100/25 µg
Number analyzed (Participants) | 39 | 42 | 39 | 44 | 81 | 83
Liters | 0.047 (0.3002) | 0.146 (0.2330) | 0.193 (0.2192) | 0.175 (0.2478) | 0.143 (0.3150) | 0.121 (0.2779)
Statistical Analysis 1: Comparison: FF 100 µg vs FF/UMEC 100/15.6 µg; Test type: Superiority or Other; p = 0.024, Final step dose response model; Mean Difference (Net) = 0.103, 95% CI 2-sided [0.014 to 0.193]
Statistical Analysis 2: Comparison: FF 100 µg vs FF/UMEC 100/62.5 µg; Test type: Superiority or Other; p = 0.024, Final step dose response model; Mean Difference (Net) = 0.103, 95% CI 2-sided [0.014 to 0.193]
Statistical Analysis 3: Comparison: FF 100 µg vs FF/UMEC 100/125 µg; Test type: Superiority or Other; p = 0.024, Final step dose response model; Mean Difference (Net) = 0.103, 95% CI 2-sided [0.014 to 0.193]
Statistical Analysis 4: Comparison: FF 100 µg vs FF/UMEC 100/250 µg; Test type: Superiority or Other; p = 0.024, Final step dose response model; Mean Difference (Net) = 0.103, 95% CI 2-sided [0.014 to 0.193]
Statistical Analysis 5: Comparison: FF 100 µg vs FF/VI 100/25 µg; Test type: Superiority or Other; p = 0.152, Final dose response model; Mean Difference (Net) = 0.073, 95% CI 2-sided [-0.027 to 0.172]

2. Secondary Outcome: Mean Change From Baseline in Rescue Medication Use at the End of Treatment Phase A
Description: All participants received the albuterol/salbutamol via MDI as a rescue medication on an as-needed basis. Total daily rescue medication use for a given day is the sum of daytime albuterol/salbutamol use recorded in PM and nighttime albuterol/salbutamol use recorded in AM the next day. The number of puffs of albuterol (salbutamol) MDI used in the last 12 hours for relief of symptoms were recorded morning and evening in the eDiary by the participants. End of Treatment Phase A is the last 7 days of Treatment Phase A. Change from Baseline at the end of Treatment Phase is the difference between the end of Treatment Phase value and the appropriate baseline week. Analysis performed using analysis of covariance with covariates of treatment, age, sex, baseline rescue medication use, pack years smoked per randomization stratification and age when first treated with an inhaler per randomization stratification. Baseline is the last 7 days of the run-in period prior to randomization
Time Frame: Baseline and End of Treatment Phase A (The end of Treatment Phase A was defined as the last 7 days of Treatment Phase A, including the AM assessments on the date of Visit 6)
Population: ITT Population. Only those participants available at the specified time point were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Puffs
Arm/Group | FF 100 µg | FF/UMEC 100/15.6 µg | FF/UMEC 100/62.5 µg | FF/UMEC 100/125 µg | FF/UMEC 100/250 µg | FF/VI 100/25 µg
Number analyzed (Participants) | 41 | 42 | 40 | 46 | 85 | 84
Puffs | 0.6 (0.29) | -0.4 (0.29) | -0.5 (0.29) | 0.0 (0.27) | -0.2 (0.21) | -0.1 (0.21)
Statistical Analysis 1: Comparison: FF 100 µg vs FF/UMEC 100/15.6 µg; Test type: Superiority or Other; p = 0.010, ANCOVA; Mean Difference (Net) = -1.0, 95% CI 2-sided [-1.7 to -0.2]
Statistical Analysis 2: Comparison: FF 100 µg vs FF/UMEC 100/62.5 µg; Test type: Superiority or Other; p = 0.004, ANCOVA; Mean Difference (Net) = -1.1, 95% CI 2-sided [-1.9 to -0.4] — Statistical analysis presented for daily rescue medication use
Statistical Analysis 3: Comparison: FF 100 µg vs FF/UMEC 100/125 µg; Test type: Superiority or Other; p = 0.083, ANCOVA; Mean Difference (Net) = -0.7, 95% CI 2-sided [-1.4 to 0.1] — Statistical analysis presented for daily rescue medication use
Statistical Analysis 4: Comparison: FF 100 µg vs FF/UMEC 100/250 µg; Test type: Superiority or Other; p = 0.014, ANCOVA; Mean Difference (Net) = -0.8, 95% CI 2-sided [-1.5 to -0.2] — Statistical analysis presented for daily rescue medication use
Statistical Analysis 5: Comparison: FF 100 µg vs FF/VI 100/25 µg; Test type: Superiority or Other; p = 0.031, ANCOVA; Mean Difference (Net) = -0.7, 95% CI 2-sided [-1.4 to -0.1] — Statistical analysis presented for daily rescue medication use

3. Secondary Outcome: Mean Change From Baseline in E-RS Total Scores at the End of Treatment Phase A
Description: A daily symptoms score for exacerbations of chronic pulmonary disease tool - Respiratory Symptoms (E-RS) is derived by summing the 11 item-level E-RS scores and has a theoretical range of 0-40, with higher values indicating more severe respiratory symptoms. The Baseline E-RS score is defined as the mean within-subject daily score over the 7 days prior to randomization, with data present for a minimum of 4 of the 7 days. Change from Baseline at the end of Treatment Phase is the difference between the end of Treatment Phase value and the appropriate Baseline week. Analysis performed using analysis of covariance with covariates of treatment, age, sex, baseline score, pack years smoked per randomization stratification and age when first treated with an inhaler per randomization stratification. Baseline is the last 7 days of the run-in period prior to randomization. All comparisons for statistical purposes are with the FF 100 µg arm.
Time Frame: as for outcome 2
Population: ITT Population. Only those participants available at the specified time point were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Score on scale
Arm/Group | FF 100 µg | FF/UMEC 100/15.6 µg | FF/UMEC 100/62.5 µg | FF/UMEC 100/125 µg | FF/UMEC 100/250 µg | FF/VI 100/25 µg
Number analyzed (Participants) | 39 | 42 | 39 | 43 | 81 | 83
Score on scale | 0.5 (0.54) | -2.6 (0.55) | -2.5 (0.56) | -1.5 (0.52) | -1.5 (0.40) | -1.1 (0.41)
Statistical Analysis 1: Comparison: FF 100 µg vs FF/UMEC 100/15.6 µg; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Net) = -3.1, 95% CI 2-sided [-4.6 to -1.7]
Statistical Analysis 2: Comparison: FF 100 µg vs FF/UMEC 100/62.5 µg; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Net) = -3.0, 95% CI 2-sided [-4.5 to -1.6]
Statistical Analysis 3: Comparison: FF 100 µg vs FF/UMEC 100/125 µg; Test type: Superiority or Other; p = 0.007, ANCOVA; Mean Difference (Net) = -2.0, 95% CI 2-sided [-3.4 to -0.6]
Statistical Analysis 4: Comparison: FF 100 µg vs FF/UMEC 100/250 µg; Test type: Superiority or Other; p = 0.002, ANCOVA; Mean Difference (Net) = -2.0, 95% CI 2-sided [-3.2 to -0.7]
Statistical Analysis 5: Comparison: FF 100 µg vs FF/VI 100/25 µg; Test type: Superiority or Other; p = 0.009, ANCOVA; Mean Difference (Net) = -1.7, 95% CI 2-sided [-2.9 to -0.4]

4. Secondary Outcome: Change From Baseline in Daily Morning (AM) PEF (Pre-dose and Pre-rescue Bronchodilator) Measured at Home and Averaged Over the Last 21 Days of Treatment Phase A
Description: Peak expiratory flow (PEF) stability limit was calculated from AM PEF measurements on the 7 days preceding Visit 3 as mean AM PEF from the available 7 days preceding Visit 3 x 80%. PEF stability limit serves as a benchmark of the participants run-in COPD status and used for comparison during the treatment phase to assess subject safety. Change from Baseline over the last 21 days of Treatment Phase A is the difference between the last 21 days of Treatment Phase A and the appropriate Baseline week. The last 21 days of Treatment Phase A include the AM assessments on the date of Visit 6. AM assessments include the date of Visit 6 and the 20 consecutive days preceding the date of Visit. Analysis performed using analysis of covariance with covariates of treatment, age, sex, Baseline AM PEF, pack years smoked per randomization stratification and age when first treated with an inhaler per randomization stratification. Baseline is the last 7 days of the run-in period prior to randomization
Time Frame: Baseline and from Day 8 through Day 29
Population: ITT Population. Only those participants available at the specified time point were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Liters per minute (L/min)
Arm/Group | FF 100 µg | FF/UMEC 100/15.6 µg | FF/UMEC 100/62.5 µg | FF/UMEC 100/125 µg | FF/UMEC 100/250 µg | FF/VI 100/25 µg
Number analyzed (Participants) | 39 | 42 | 39 | 43 | 81 | 83
Liters per minute (L/min) | -14.2 (4.62) | 3.9 (4.70) | 7.6 (4.76) | 5.5 (4.40) | 10.5 (3.37) | 4.3 (3.47)
Statistical Analysis 1: Comparison: FF 100 µg vs FF/UMEC 100/15.6 µg; Test type: Superiority or Other; p = 0.004, ANCOVA; Mean Difference (Net) = 18.1, 95% CI [5.9 to 30.3]
Statistical Analysis 2: Comparison: FF 100 µg vs FF/UMEC 100/62.5 µg; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Net) = 21.8, 95% CI 2-sided [9.4 to 34.1]
Statistical Analysis 3: Comparison: FF 100 µg vs FF/UMEC 100/125 µg; Test type: Superiority or Other; p = 0.001, ANCOVA; Mean Difference (Net) = 19.7, 95% CI 2-sided [7.7 to 31.7]
Statistical Analysis 4: Comparison: FF 100 µg vs FF/UMEC 100/250 µg; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Net) = 24.8, 95% CI 2-sided [14.1 to 35.4]
Statistical Analysis 5: Comparison: FF 100 µg vs FF/VI 100/25 µg; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Net) = 18.5, 95% CI 2-sided [8.0 to 29.1]

5. Secondary Outcome: Change From Trough in Clinic Forced Expiratory Volume (FEV1) at 3 Hours Post-study Treatment at Visit 5/Day 28
Description: FEV1 was measured in the morning by spirometry. At Visit 5, after trough FEV1 is measured, subject received investigational product. 3 hours post-dose, spirometry was repeated and subject then received 2 puffs of albuterol/salbutamol. After 30 minutes,spirometry was repeated.. Change from Baseline in clinic trough (pre-dose) FEV1 is the difference in the trough value at 3 hours post-dose peak FEV1 and the Baseline value. If the trough value or the Baseline was missing, then change from Baseline was considered as missing. Baseline value of clinic FEV1 is the last acceptable/borderline acceptable (pre-dose) FEV1 value obtained prior to randomization (from Visit 3 pre-dose or from Visit 2 pre-bronchodilator). Analysis done using analysis of covariance with covariates of treatment, age, sex, baseline clinic trough FEV1, pre-dose trough FEV1 at Visit 5, pack years smoked per randomization stratification and age when first treated with an inhaler per randomization stratification.
Time Frame: Baseline and Day 28
Population: ITT Population. Only those participants available at the specified time point were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Liters (L)
Arm/Group | FF 100 µg | FF/UMEC 100/15.6 µg | FF/UMEC 100/62.5 µg | FF/UMEC 100/125 µg | FF/UMEC 100/250 µg | FF/VI 100/25 µg
Number analyzed (Participants) | 38 | 42 | 39 | 45 | 81 | 82
Liters (L) | 0.048 (0.0307) | 0.093 (0.0305) | 0.088 (0.0309) | 0.072 (0.0279) | 0.052 (0.0220) | 0.124 (0.0227)
Statistical Analysis 1: Comparison: FF 100 µg vs FF/UMEC 100/15.6 µg; Test type: Superiority or Other; p = 0.264, ANCOVA; Mean Difference (Net) = 0.045, 95% CI 2-sided [-0.034 to 0.125]
Statistical Analysis 2: Comparison: FF 100 µg vs FF/UMEC 100/62.5 µg; Test type: Superiority or Other; p = 0.328, ANCOVA; Mean Difference (Net) = 0.040, 95% CI 2-sided [-0.041 to 0.121]
Statistical Analysis 3: Comparison: FF 100 µg vs FF/UMEC 100/125 µg; Test type: Superiority or Other; p = 0.534, ANCOVA; Mean Difference (Net) = 0.025, 95% CI 2-sided [-0.054 to 0.103]
Statistical Analysis 4: Comparison: FF 100 µg vs FF/UMEC 100/250 µg; Test type: Superiority or Other; p = 0.895, ANCOVA; Mean Difference (Net) = 0.005, 95% CI 2-sided [-0.065 to 0.075]
Statistical Analysis 5: Comparison: FF 100 µg vs FF/VI 100/25 µg; Test type: Superiority or Other; p = 0.031, ANCOVA; Mean Difference (Net) = 0.076, 95% CI 2-sided [0.007 to 0.146]

6. Secondary Outcome: Change in Clinic FEV1 Following 2 Puffs of Albuterol/Salbutamol Given 3 Hours Post-study Treatment Dose at Visit 5/Day 28
Description: FEV1 is defined as forced expiratory volume in one second and measured in the morning at Visits 1 through 8 between 6:00 and 11:00 electronically by spirometry. Reversibility was measured at Visit 1 and Visit 2 for study eligibility by change in clinic FEV1 within 20 to 60 minutes following 4 inhalations of albuterol/salbutamol and again measured 3 hours after dosing at Visit 5 by change in clinic FEV1 30 minutes following 2 inhalations of albuterol/salbutamol. Baseline value of clinic FEV1 is the last acceptable/borderline acceptable (pre-dose) FEV1 value obtained prior to randomization (either from Visit 3 pre-dose or from Visit 2 pre-bronchodilator). Analysis performed using analysis of covariance with covariates of treatment, age, sex, baseline clinic trough FEV1, pre-albuterol/salbutamol FEV1 at Visit 5, pack years smoked per randomization stratification and age when first treated with an inhaler per randomization stratification.
Time Frame: Baseline and Day 28
Population: ITT Population. Only those participants available at the specified time point were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Liters (L)
Arm/Group | FF 100 µg | FF/UMEC 100/15.6 µg | FF/UMEC 100/62.5 µg | FF/UMEC 100/125 µg | FF/UMEC 100/250 µg | FF/VI 100/25 µg
Number analyzed (Participants) | 37 | 40 | 38 | 42 | 80 | 80
Liters (L) | 0.249 (0.0287) | 0.161 (0.0284) | 0.159 (0.0284) | 0.160 (0.0262) | 0.189 (0.0202) | 0.087 (0.0209)
Statistical Analysis 1: Comparison: FF 100 µg vs FF/UMEC 100/15.6 µg; Test type: Superiority or Other; p = 0.019, ANCOVA; Mean Difference (Net) = -0.088, 95% CI 2-sided [-0.162 to -0.014]
Statistical Analysis 2: Comparison: FF 100 µg vs FF/UMEC 100/62.5 µg; Test type: Superiority or Other; p = 0.017, ANCOVA; Mean Difference (Net) = -0.091, 95% CI 2-sided [-0.165 to -0.016]
Statistical Analysis 3: Comparison: FF 100 µg vs FF/UMEC 100/125 µg; Test type: Superiority or Other; p = 0.017, ANCOVA; Mean Difference (Net) = -0.089, 95% CI 2-sided [-0.162 to -0.016]
Statistical Analysis 4: Comparison: FF 100 µg vs FF/UMEC 100/250 µg; Test type: Superiority or Other; p = 0.066, ANCOVA; Mean Difference (Net) = -0.060, 95% CI 2-sided [-0.124 to 0.004]
Statistical Analysis 5: Comparison: FF 100 µg vs FF/VI 100/25 µg; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Net) = -0.163, 95% CI 2-sided [-0.227 to -0.099]

ADVERSE EVENTS:
Time Frame: AEs and SAEs were collected from start of the run-in period until follow-up (Visit 8 + 7 days (+/- 2 days). SAEs related to participation or GSK concomitant medication were recorded from time of consent up to and including any follow up contact.
Description: AEs and SAEs were collected for the ITT population, comprised of all participants randomized to treatment who received at least one dose of randomized study medication in the treatment period. Assessed as related to participation might include; study treatment, protocol-mandated procedures, invasive tests, or change in existing therapy.
Arm/Group | FF 100 µg | FF/UMEC 100/15.6 µg | FF/UMEC 100/62.5 µg | FF/UMEC 100/125 µg | FF/UMEC 100/250 µg | FF/VI 100/25 µg | FF/UMEC/VI 100/250/25 µg
Serious Adverse Events (participants affected / at risk) | 0/111 | 0/42 | 0/40 | 0/46 | 1/210 | 0/146 | 0/163
Other Adverse Events (participants affected / at risk) | 6/111 | 5/42 | 4/40 | 4/46 | 5/210 | 4/146 | 0/163
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FF 100 µg (N=111) | FF/UMEC 100/15.6 µg (N=42) | FF/UMEC 100/62.5 µg (N=40) | FF/UMEC 100/125 µg (N=46) | FF/UMEC 100/250 µg (N=210) | FF/VI 100/25 µg (N=146) | FF/UMEC/VI 100/250/25 µg (N=163)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — One subject had a non-fatal SAE of pneumonia 2 days after withdrawal, which resolved. This subject also had 2 fatal SAEs; TIA and PE, onset 14 and 17 days after last dose, respectively. The investigator considered pneumonia and PE treatment-related.
Transient ischaemic attack (TIA) (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (PE) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FF 100 µg (N=111) | FF/UMEC 100/15.6 µg (N=42) | FF/UMEC 100/62.5 µg (N=40) | FF/UMEC 100/125 µg (N=46) | FF/UMEC 100/250 µg (N=210) | FF/VI 100/25 µg (N=146) | FF/UMEC/VI 100/250/25 µg (N=163)
Toothache (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 6 (6) | 3 (3) | 2 (3) | 2 (2) | 4 (4) | 4 (4) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.